CLINICAL TRIAL: NCT03926507
Title: Study of F18 Fluciclovine PET CT for Assessment of Glioblastoma Tumor Volume and Radiation Response
Brief Title: F18 Fluciclovine PET/CT in Assessing Tumor Volume and Radiation Therapy Response in Patients With Glioblastoma Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0869; NCI-2019-01532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0869 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — fluciclovine F-18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (fluciclovine F18 PET/CT) (Experimental): Patients receive fluciclovine F18 IV and undergo 4 PET/CT scans over 10 minutes paired with standard of care MRI within 14 days prior to initial maximal tumor resection, within 7 days prior to initiation of radiation therapy, 28 days after the completion of radiation therapy, and 6 months after the completion of radiation therapy.
  Interventions: Procedure: Computed Tomography; Other: Fluciclovine F18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Other: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This early phase I trial studies how well F18 fluciclovine positron emission tomography (PET)/computed tomography (CT) works in assessing tumor volume and radiation therapy response in patients with glioblastoma undergoing surgery. Radioactive imaging agents, such as F18 fluciclovine, used during PET/CT scan may help measure tumor size compared to standard of care magnetic resonance imaging (MRI) contrast agents in patients receiving radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare fluciclovine F18 (F18 fluciclovine) PET CT for tumor volume assessment compared to T2 fluid attenuated inversion recovery (FLAIR) and T1 post contrast magnetic resonance (MR) brain imaging.

SECONDARY OBJECTIVES:

I. To assess changes in F18 fluciclovine defined disease with surgery and radiation.

II. To assess the relationship between post-radiation enhancing brain tissue and F18 fluciclovine activity.

EXPLORATORY OBJECTIVES:

I. To assess the association between results from pathology and F18 fluciclovine, T2 FLAIR, and T1 post-contrast MR brain imaging.

OUTLINE:

Patients receive fluciclovine F18 intravenously (IV) and undergo 4 PET/CT scans over 10 minutes paired with standard of care MRI within 14 days prior to initial maximal tumor resection, within 7 days prior to initiation of radiation therapy, 28 days after the completion of radiation therapy, and 6 months after the completion of radiation therapy.

After completion of study, patients will be followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for brain tumor resection and radiation with lesion suspected to be or previously biopsy proven to be a glioblastoma.
* Patient is able to understand and give consent to participation in the study.

Exclusion Criteria:

* Pregnant.
* Known allergy to gadolinium-based contrast agents or F18 fluciclovine.
* Renal failure as evidenced by a glomerular filtration rate (GFR) of less than 60 mL/min/1.73 m^2.
* Pacemakers, electronic stimulation, metallic foreign bodies and devices and/or other conditions that are not MR safe, which include but are not limited to:

  * Electronically, magnetically, and mechanically activated implants
  * Ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators and cardiac pacemakers
  * Metallic splinters in the eye
  * Ferromagnetic hemostatic clips in the central nervous system (CNS) or body
  * Cochlear implants
  * Other pacemakers, e.g., for the carotid sinus
  * Insulin pumps and nerve stimulators
  * Non-MR safe lead wires
  * Prosthetic heart valves (if dehiscence is suspected)
  * Non-ferromagnetic stapedial implants
  * Pregnancy
  * Claustrophobia that does not readily respond to oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Tumor volume | Up to 6 months
  Will be assessed with fluciclovine F18 (F18 fluciclovine) positron emission tomography (PET) computed tomography (CT). The three volumes measured (amino acid hypermetabolic volume [AHV], T2 fluid attenuated inversion recovery [FLAIR] and T1 contrast [T1C]) will be compared to each other for each patient, and plotted as boxplots, both raw (as mL) and as normalized values (to the T1C volume) to facilitate comparisons between patients.

SECONDARY OUTCOMES:
Changes in F18 fluciclovine defined disease with surgery and radiation | Baseline up to 6 months
  Will compare tumor volumes measured by this method between the initial time point and the three follow-up time points within patients using Wilcoxon rank-sum tests.
Post-radiation enhancing brain tissue | Up to 6 months
  To assess the relationship between post-radiation enhancing brain tissue and F18 fluciclovine activity, will use rank correlation analysis.

OTHER OUTCOMES:
Results from pathology | Up to 6 months
  Will use rank correlation analysis to assess the association between results from pathology and F18 fluciclovine, T2 FLAIR, and T1 post-contrast MR brain imaging. The association between tumor histology (glioma/non-glioma) and grade and tumor volumes from imaging results will be assessed using Wilcoxon rank-sum tests and rank correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Johnson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03926507/ICF_000.pdf